CLINICAL TRIAL: NCT06024343
Title: Long-term Outcome in Minimally Invasive Pancreatic Enucleation With Main Pancreatic Duct Exposure, Repair or Reconstruction: A Prospective Cohort Study
Brief Title: Minimally Invasive Pancreatic Enucleation With Main Pancreatic Duct Exposure, Repair or Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Fudan University Shanghai Cancer Center, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPAC-MIEN-1
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Pancreatic Tumor, Benign; Pancreatic Neuroendocrine Tumor; Solid Pseudopapillary Tumor of the Pancreas
Keywords: Pancreatic benign or low-grade malignant tumors; Minimally invasive enucleation; Main Pancreatic Duct Repair or Reconstruction; Long-term prognosis; Quality of life
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoma, Islet Cell | interventions — Wound Healing; Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPD Manipulation (Experimental): During laparoscopic or robotic pancreatic tumor enucleation, tumors located near or surrounding the main pancreatic duct (MPD) can result in the exposure, injury, or transection of the MPD, requiring MPD repair and reconstruction.
  Interventions: Procedure: MPD Exposure, Repair or Reconstruction
- MPD not exposed (No Intervention): In laparoscopic or robotic pancreatic tumor enucleation procedures where the MPD remains unexposed, there is no need for MPD repair and reconstruction.

INTERVENTIONS:
Procedure: MPD Exposure, Repair or Reconstruction — During laparoscopic or robotic pancreatic tumor enucleation, if the main pancreatic duct (MPD) is injured due to its proximity or encasement by the tumor, MPD manipulation is performed. MPD manipulation is categorized into three scenarios: exposed but not injured; simple suture repair (using 5-0/6-0 PROLENE polypropylene suture); and suture repair/reconstruction following stent insertion. Using the F6 ventricular drainage catheter with 1-2 side holes trimmed as the stent, typically requiring 10 cm for passage through the duodenal papilla and 3-4 cm if not passing through. Following stent placement, intermittent suturing reconstructs the MPD, with one stitch securing the stent by passing through both the stent side wall and the MPD.
  Arms: MPD Manipulation

SUMMARY:
The aim of this study is to evaluate the impact of concomitant main pancreatic duct exposure, repair, or reconstruction during minimally invasive pancreatic tumor enucleation on long-term patient prognosis and quality of life.

DETAILED DESCRIPTION:
Standard surgical procedures for benign or low-grade malignant pancreatic tumors is associated with increased risks of postoperative complications and long-term pancreatic functional impairment, while parenchyma-sparing pancreatectomy such as enucleation can reduce the incidence of complications and preserve healthy parenchyma, thereby preserve both endocrine and exocrine pancreatic function. It has been reported that pancreatic tumor enucleation is a safe and feasible approach in preserving normal physiological function in patients undergoing pancreatic surgery.

With the growing emphasis on routine screenings and the application of high-quality thin-slice imaging techniques, the detection rates of pancreatic tumors have witnessed a steady increase. Additionally, there is a notable trend towards younger patients being diagnosed with pancreatic tumors. Consequently, in conjunction with ensuring safe and thorough tumor resection while maximizing preservation of pancreatic function, there is a current clinical demand to further reduce surgical trauma.

Literature reviews and meta-analyses have demonstrated that minimally invasive enucleation procedures offer well-known advantages associated with minimally invasive approaches, such as shorter postoperative hospital stays and lower overall complication rates. While the occurrence rate of severe complications, such as postoperative hemorrhage, remains relatively low, the development of postoperative pancreatic fistula (POPF) continues to pose a challenging issue.

The distance between the tumor and the main pancreatic duct (MPD) is considered a crucial factor influencing the occurrence of POPF after enucleation. However, these data have been rarely described in previous studies, making it challenging to accurately assess their actual impact on the rate of POPF occurrence. Heeger et al. suggested that the risk of POPF increases with closer proximity of the tumor to the MPD. The incidence of POPF was higher in deep-seated tumors after pancreatic enucleation (distance to MPD <3 mm) compared to superficial tumors (>3 mm) (73.3% vs. 30.0%, P=0.002). Other studies have even limited this critical distance to 2mm. Some research has indicated that if the tumor invades or encases the MPD, enucleation surgery should be contraindicated, and standard resection should be preferred to avoid the risk of POPF postoperatively. However, a retrospective analysis by Strobel et al. on 166 cases of pancreatic tumor enucleation demonstrated that even tumors in close proximity to the MPD can be safely resected, although their study did not include cases with tumor encasement of the MPD.

During the expansive growth of solid tumors such as neuroendocrine tumors and solid pseudopapillary neoplasms, they can compress the MPD, causing inflammatory adhesions. Cystic tumors can also surround the MPD as they grow. Enucleation of these tumors may inevitably lead to exposure, injury, or transection of the MPD, necessitating repair and reconstruction. Recent years have seen successful cases reported of end-to-end anastomosis of the MPD. Minimally invasive techniques have also facilitated the promotion of MPD repair or bridging reconstruction surgeries. However, there remains a lack of comprehensive research data in this field.

The safety and feasibility of minimally invasive pancreatic tumor enucleation procedures involving MPD exposure, repair, or reconstruction, the control of POPF, and the long-term prognosis and quality of life of patients after MPD repair or reconstruction remain unclear. Therefore, this study aims to conduct a prospective cohort study. The results of this study will serve as a valuable reference for clinical practice and promote the development and application of minimally invasive pancreatic tumor enucleation procedures.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 75 years, regardless of gender;
2. patients with solitary benign or low-grade malignant pancreatic tumors, including NET, SPN, and cystic tumors;
3. eligible for pancreatic parenchyma-sparing resection (PSR) according to contemporary guidelines;
4. patients with an ECOG performance status of 0 or 1;
5. successfully received MIEN (laparoscopic or robotic)

Exclusion Criteria:

1. body mass index > 35 kg/m2;
2. concomitant malignancies;
3. intraoperative frozen section or postoperative pathology indicating malignancy, requiring conversion to oncologic resection;
4. loss to follow-up within 90 days postoperatively.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Clinically Relevant Postoperative Pancreatic Fistula | Within 90 days after surgery.
  Clinically Relevant Pancreatic Fistula including Grade B fistulas, which require treatment beyond simple drainage, as well as Grade C fistulas.

SECONDARY OUTCOMES:
Perioperative complication rate according to the Clavien-Dindo classification | Within 90 days after surgery.
  Adverse events that occur during or after the surgery, reported according to the Clavien-Dindo classification.
Postoperative pancreatic hemorrhage (PPH) rate | Within 90 days after surgery.
  Postoperative pancreatic hemorrhage (PPH) rate within 90 days after surgery, reported according to the ISGPS definition.
Delayed gastric emptying (DGE) rate | Within 90 days after surgery.
  Delayed gastric emptying (DGE) rate within 90 days after surgery, reported according to the ISGPS definition.
Reoperation rate | Within 90 days after surgery.
  Reoperation rate within 90 days after surgery.
Rate of pancreatic enzyme-dependent malabsorption | Through study completion, an average of 3 year.
  Postoperative pancreatic enzyme-dependent malabsorption rate.
Rate of new-onset diabetes | Through study completion, an average of 3 year.
  Postoperative new-onset diabetes rate.
Life quality satisfaction evaluated according to EORTC C30 scale | Through study completion, an average of 3 year.
  The patient's health-related quality of life after surgical intervention. It includes physical, emotional, and social aspects of a patient's well-being. This study evaluated quality of life using a telephone survey and the EORTC C30 scales.
R0 resection rate | From the date of surgery to 1 month after surgery.
  R0 margin rate on postoperative pathological assessment.
Recurrence-free survival (RFS) | Through study completion, an average of 3 year.
  The time of surgery to the time of tumor recurrence or death.

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun Yu, MD, PhD, Principal Investigator — Fudan University; Xiaowu Xu, MD, Study Director — Fudan University
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cauley CE, Pitt HA, Ziegler KM, Nakeeb A, Schmidt CM, Zyromski NJ, House MG, Lillemoe KD. Pancreatic enucleation: improved outcomes compared to resection. J Gastrointest Surg. 2012 Jul;16(7):1347-53. doi: 10.1007/s11605-012-1893-7. Epub 2012 Apr 24. PMID 22528577
- [Background] Giuliani T, De Pastena M, Paiella S, Marchegiani G, Landoni L, Festini M, Ramera M, Marinelli V, Casetti L, Esposito A, Bassi C, Salvia R. Pancreatic Enucleation Patients Share the Same Quality of Life as the General Population at Long-Term Follow-Up: A Propensity Score-Matched Analysis. Ann Surg. 2023 Mar 1;277(3):e609-e616. doi: 10.1097/SLA.0000000000004911. Epub 2021 Apr 14. PMID 33856383
- [Background] Kromrey ML, Bulow R, Hubner J, Paperlein C, Lerch MM, Ittermann T, Volzke H, Mayerle J, Kuhn JP. Prospective study on the incidence, prevalence and 5-year pancreatic-related mortality of pancreatic cysts in a population-based study. Gut. 2018 Jan;67(1):138-145. doi: 10.1136/gutjnl-2016-313127. Epub 2017 Sep 6. PMID 28877981
- [Background] van Huijgevoort NCM, Del Chiaro M, Wolfgang CL, van Hooft JE, Besselink MG. Diagnosis and management of pancreatic cystic neoplasms: current evidence and guidelines. Nat Rev Gastroenterol Hepatol. 2019 Nov;16(11):676-689. doi: 10.1038/s41575-019-0195-x. Epub 2019 Sep 16. PMID 31527862
- [Background] Dasari A, Shen C, Halperin D, Zhao B, Zhou S, Xu Y, Shih T, Yao JC. Trends in the Incidence, Prevalence, and Survival Outcomes in Patients With Neuroendocrine Tumors in the United States. JAMA Oncol. 2017 Oct 1;3(10):1335-1342. doi: 10.1001/jamaoncol.2017.0589. PMID 28448665
- [Background] Zhou Y, Zhao M, Wu L, Ye F, Si X. Short- and long-term outcomes after enucleation of pancreatic tumors: An evidence-based assessment. Pancreatology. 2016 Nov-Dec;16(6):1092-1098. doi: 10.1016/j.pan.2016.07.006. Epub 2016 Jul 9. PMID 27423534
- [Background] Guerra F, Giuliani G, Bencini L, Bianchi PP, Coratti A. Minimally invasive versus open pancreatic enucleation. Systematic review and meta-analysis of surgical outcomes. J Surg Oncol. 2018 Jun;117(7):1509-1516. doi: 10.1002/jso.25026. Epub 2018 Mar 25. PMID 29574729
- [Background] Dalla Valle R, Cremaschi E, Lamecchi L, Guerini F, Rosso E, Iaria M. Open and minimally invasive pancreatic neoplasms enucleation: a systematic review. Surg Endosc. 2019 Oct;33(10):3192-3199. doi: 10.1007/s00464-019-06967-9. Epub 2019 Jul 30. PMID 31363894
- [Background] Shukla PJ, Barreto SG, Shrikhande SV. Enucleation of pancreatic neoplasms (Br J Surg 2007; 94: 1254-1259). Br J Surg. 2008 Feb;95(2):261; author reply 261-2. doi: 10.1002/bjs.6148. No abstract available. PMID 18196559
- [Background] Brient C, Regenet N, Sulpice L, Brunaud L, Mucci-Hennekine S, Carrere N, Milin J, Ayav A, Pradere B, Hamy A, Bresler L, Meunier B, Mirallie E. Risk factors for postoperative pancreatic fistulization subsequent to enucleation. J Gastrointest Surg. 2012 Oct;16(10):1883-7. doi: 10.1007/s11605-012-1971-x. Epub 2012 Aug 8. PMID 22872510
- [Background] Bartolini I, Bencini L, Bernini M, Farsi M, Calistri M, Annecchiarico M, Moraldi L, Coratti A. Robotic enucleations of pancreatic benign or low-grade malignant tumors: preliminary results and comparison with robotic demolitive resections. Surg Endosc. 2019 Sep;33(9):2834-2842. doi: 10.1007/s00464-018-6576-3. Epub 2018 Nov 12. PMID 30421079
- [Background] Ei S, Mihaljevic AL, Kulu Y, Kaiser J, Hinz U, Buchler MW, Hackert T. Enucleation for benign or borderline tumors of the pancreas: comparing open and minimally invasive surgery. HPB (Oxford). 2021 Jun;23(6):921-926. doi: 10.1016/j.hpb.2020.10.001. Epub 2020 Oct 18. PMID 33087306
- [Background] Zhang RC, Zhou YC, Mou YP, Huang CJ, Jin WW, Yan JF, Wang YX, Liao Y. Laparoscopic versus open enucleation for pancreatic neoplasms: clinical outcomes and pancreatic function analysis. Surg Endosc. 2016 Jul;30(7):2657-65. doi: 10.1007/s00464-015-4538-6. Epub 2015 Oct 20. PMID 26487211
- [Background] Strobel O, Cherrez A, Hinz U, Mayer P, Kaiser J, Fritz S, Schneider L, Klauss M, Buchler MW, Hackert T. Risk of pancreatic fistula after enucleation of pancreatic tumours. Br J Surg. 2015 Sep;102(10):1258-66. doi: 10.1002/bjs.9843. Epub 2015 Jun 24. PMID 26109380
- See also: In 2021, Professor Liu Rong and colleagues introduced the concept of pancreatic duct surgery for the first time and outlined four main surgical approaches. — https://doi.org/10.1016/j.isurg.2022.11.001